CLINICAL TRIAL: NCT05003908
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Diabetes
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of efficacy
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-10-ATG-11-01
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
Keywords: Diabetes; stem cell treatment
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Diabetes

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Diabetes. Patients with Diabetes will receive a single intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease requiring chemotherapeutic drugs such as methotrexate, an autologous T Cell vaccine will be utilized created from the patient's own T cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: the level of A1C | Four year follow-up
  A1C blood test will be completed for each follow up point.
Efficacy: the level of C-Peptide | Four year follow-up
  C-Peptide test will be completed for each follow up point.
Efficacy: Insulin dose reduction | Four year follow-up
  Changes of insulin dosage for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

REFERENCES:
- [Background] Hu J, Yu X, Wang Z, Wang F, Wang L, Gao H, Chen Y, Zhao W, Jia Z, Yan S, Wang Y. Long term effects of the implantation of Wharton's jelly-derived mesenchymal stem cells from the umbilical cord for newly-onset type 1 diabetes mellitus. Endocr J. 2013;60(3):347-57. doi: 10.1507/endocrj.ej12-0343. Epub 2012 Nov 16. PMID 23154532
- [Background] Jiang R, Han Z, Zhuo G, Qu X, Li X, Wang X, Shao Y, Yang S, Han ZC. Transplantation of placenta-derived mesenchymal stem cells in type 2 diabetes: a pilot study. Front Med. 2011 Mar;5(1):94-100. doi: 10.1007/s11684-011-0116-z. Epub 2011 Mar 17. PMID 21681681
- [Background] Cai J, Wu Z, Xu X, Liao L, Chen J, Huang L, Wu W, Luo F, Wu C, Pugliese A, Pileggi A, Ricordi C, Tan J. Umbilical Cord Mesenchymal Stromal Cell With Autologous Bone Marrow Cell Transplantation in Established Type 1 Diabetes: A Pilot Randomized Controlled Open-Label Clinical Study to Assess Safety and Impact on Insulin Secretion. Diabetes Care. 2016 Jan;39(1):149-57. doi: 10.2337/dc15-0171. Epub 2015 Dec 1. PMID 26628416